CLINICAL TRIAL: NCT03462160
Title: Effectiveness of Prophylaxis of Urinary Tract Infections in Children With a Probiotic Containing Lactobacillus Rhamnosus PL1 and Lactobacillus Plantarum PM1, a Randomised Clinical Trial
Brief Title: Effectiveness of Probiotics Prophylaxis of Urinary Tract Infections in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Miralex Sp. z o.o. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UTI probiotic
Record Dates: First submitted 2018-02-28; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Prevention of Urinary Tract Infections in Children
Keywords: Urinary Tract Infection; prophylaxis; probiotics
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo supply for 90 days (Placebo Comparator): Patients will receive placebo (in blinded sachets)
  Interventions: Other: Placebo control group
- Probiotic supply for 90 days (Experimental): Patients will receive probiotics containing Lactobacillus rhamnosus PL1 and Lactobacillus plantarum PM1 (in blinded sachets).
  Interventions: Dietary Supplement: Probiotic experimental group

INTERVENTIONS:
Other: Placebo control group — Placebo will be administered orally, after dissolving the sachet in lukewarm water, every evening during the meal. The placebo appearance will be similar to the probiotic.
  Arms: Placebo supply for 90 days
Dietary Supplement: Probiotic experimental group — Probiotic UroLact containing Lactobacillus rhamnosus PL1 and Lactobacillus plantarum PM1 will be administered orally, after dissolving the sachet in lukewarm water, every evening during the meal.
  Arms: Probiotic supply for 90 days

SUMMARY:
The investigators aim to assess the effectiveness of prophylaxis of urinary tract infections in children with a probiotic containing Lactobacillus rhamnosus PL1 and Lactobacillus plantarum PM1. It is formulated a hypothesis that a 3-months course of probiotic prophylasis is more effective than placebo.

DETAILED DESCRIPTION:
In previously published European and global guidelines, there has been no consensus among experts regarding the prophylaxis of recurrence urinary tract infections. Depending on the recommendation, the prevention of recurrence UTI should be used, not justified, or should be used in special cases. However, preparations that will be effective in preventing UTI and will not cause bacterial resistance are still sought.

106 patients aged 3 to 18 years with recurrence UTIs (defined as: ≥2 infections in the upper urinary tract or 1 UTI in the upper urinary tract and ≥1 in the lower urinary tract or ≥3 or more UTI in the lower urinary tract in one year) or children with ≥1 infection in the upper urinary tract and ≥1 of recurrent UTIs risk factors (congenital anomalies of the kidney and urinary tract, constipation, bladder dysfunction, myelomeningocele, sexual activity in girls) will be randomly assigned to receive a 90-days prophylaxsis arm (probiotic UroLact containing Lactobacillus Rhamnosus PL1 and Lactobacillus Plantarum PM1) or a 90-days placebo arms.

The primary outcome measure will be frequencies of recurrence of UTI during the 6 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* recurrent UTIs (defined as: ≥2 infections in the upper urinary tract or 1 UTI in the upper urinary tract and ≥1 in the lower urinary tract or ≥3 or more UTI in the lower urinary tract in one year) OR 1 infection in the upper urinary tract and ≥1 of recurrent UTIs risk factors: congenital anomalies of the kidney and urinary tract, constipation, bladder dysfunction, myelomeningocele, sexual activity in girls
* ≥1 episode of urinary tract infection in the last 6 months

Exclusion Criteria:

* intake of probiotic preparations for ≥1 month in the last 3 months
* known allergy to the study products
* immunosuppression therapy
* disease with immune deficiency
* children with other coexisting infection, e.g. meningitis, sepsis, pneumonia, otitis

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
frequencies of recurrence of UTI | 6 months after intervention
  New onset of symptomatic UTI within the 6 months follow-up period.

SECONDARY OUTCOMES:
frequencies of hospitalization due to UTI | 6 months after intervention
the number of days of antibiotic therapy due to UTI | 6 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Panczyk-Tomaszewska, Assistant Professor, Study Chair — Medical University of Warsaw; Maria Daniel, MD, Principal Investigator — Medical University of Warsaw; Hanna Szymanik-Grzelak, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Children's Hospital for The Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tewary K, Narchi H. Recurrent urinary tract infections in children: Preventive interventions other than prophylactic antibiotics. World J Methodol. 2015 Jun 26;5(2):13-9. doi: 10.5662/wjm.v5.i2.13. eCollection 2015 Jun 26. PMID 26140267
- [Result] Schwenger EM, Tejani AM, Loewen PS. Probiotics for preventing urinary tract infections in adults and children. Cochrane Database Syst Rev. 2015 Dec 23;2015(12):CD008772. doi: 10.1002/14651858.CD008772.pub2. PMID 26695595
- [Result] Hosseini M, Yousefifard M, Ataei N, Oraii A, Mirzay Razaz J, Izadi A. The efficacy of probiotics in prevention of urinary tract infection in children: A systematic review and meta-analysis. J Pediatr Urol. 2017 Dec;13(6):581-591. doi: 10.1016/j.jpurol.2017.08.018. Epub 2017 Oct 9. PMID 29102297
- [Derived] Daniel M, Szymanik-Grzelak H, Turczyn A, Panczyk-Tomaszewska M. Lactobacillus rhamnosus PL1 and Lactobacillus plantarum PM1 versus placebo as a prophylaxis for recurrence urinary tract infections in children: a study protocol for a randomised controlled trial. BMC Urol. 2020 Oct 23;20(1):168. doi: 10.1186/s12894-020-00723-1. PMID 33097017